CLINICAL TRIAL: NCT05093166
Title: Prospective, Open-label, Uncontrolled Pilot Clinical Trial to Assess the Safety and Efficacy of Autologous Cultured Oral Mucosa Grafts for Urethral Reconstruction in Patients Due to Hypospadias Treatment Failure
Brief Title: Clinical Trial to Assess the Safety and Efficacy of Investigational Product in Patients Due to Hypospadias Treatment Failure
Acronym: HOLOUR
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the current re-organization at the Sponsor site
Sponsor: Holostem s.r.l. (Industry)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); University of Modena and Reggio Emilia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTA-HUR-01
Record Dates: First submitted 2021-09-03; First posted 2021-10-26 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Hypospadias
Keywords: Hypospadias treatment failure; Urethral reconstruction; Cell therapy; Stem cells
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urethral reduced functionality and/or lesions due to previous hypospadias treatment failure (Experimental): The first step consists in a small oral mucosa biopsy collection by surgeon under general anaesthesia. The biopsy will be processed in a laboratory of a regenerative medicine manufacturing site where the epithelial cells will be isolated, expanded and prepared as final graft to be implanted.
  The treatment for urethra reconstruction required a two stage urethroplasty:
  1. First stage: application of Holour on the wound bed prepared according to standard surgery The penis will be immobilized for some days after this operation.
  2. Second stage: surgical procedure for urethral tubularization and penile reconstruction according to standard surgical procedure.
  The surgical procedures may be followed by a post-implantation treatment (if necessary) with corticosteroids and antibiotics.
  Interventions: Drug: "Ex vivo" expanded autologous human oral epithelium containing stem cells

INTERVENTIONS:
Drug: "Ex vivo" expanded autologous human oral epithelium containing stem cells — The treatment includes a single administration of investigational product through a dedicated surgical procedure of penis wound bed preparation, epithelial surface adaption and product application followed by urethra tubularization and penis reconstruction.

SUMMARY:
The purpose of this trial is to assess the safety and efficacy of Holour in patients suffering from hypospadias treatment failure. Holour is intended for urethral replacement and is made from ex vivo expanded autologous oral mucosal cells including stem cells.

DETAILED DESCRIPTION:
Holour is a prospective, open-label, uncontrolled pilot clinical trial phase i/ii. The aim of this clinical trial is to perform a tissue engineering therapy to assess the safety (at 3 and 12 months) and efficacy (at 12 months) of the autologous treatment.

Patients will be screened according to the study inclusion and exclusion criteria and will be candidate for the treatment if all eligibility criteria are met. Up to 8 patients will be treated by means of autologous cultured oral mucosa grafts containing oral mucosa stem cells. Holour is produced by ex vivo expansion of cells obtained from oral mucosa biopsy collected from patient. The biopsy will be processed in a laboratory of a regenerative medicine manufacturing site where the epithelial cells will be isolated, expanded and prepared as final graft to be implanted. Holour administration will be planned according to the procedures and the need of the patient.

The entire procedure envisages the following steps:

1. Oral mucosa biopsy to manufacture autologous grafts of Holour.
2. Penile urethroplasty in two stages:

   * First stage: application of holour on the wound bed prepared according to standard surgery.
   * Second stage: penis reconstruction according to standard surgical procedure. The surgical procedures may be followed by a post-implantation treatment (if necessary) with corticosteroids and antibiotics.

The treatment includes a single administration of Holour; in case of "failure" of the first procedure eligible patients can undergo to a second implantation.

Three months after the transplantation, primary endpoint will be evaluated by the investigator. The study completion will be reached when 1 year (secondary endpoint) of follow-up after the last transplant in the last patient will be accomplished.

The end of the trial is defined as the last visit of the last patient after the last treatment if any.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent prior to any study-related procedures (Caregivers); Patients whose parents/legal representatives have been thoroughly informed of the aim of the study procedures and provided signed and dated written informed consent;
2. Male patients between 5 and 17 years old (less than 18 years old);
3. Need for urethroplasty in failed hypospadias treatment;
4. Hypospadias complications shown by clinical evaluation, uroflowmetry with post-micturition residual evaluation and/or retrograde urethrography and/or urethroscopy;
5. Uroflowmetry rate: Uroflowmetry with a plateau-shaped curve and low qmax according to paediatric uroflow normograms;
6. Absence of other contraindications to HOLOUR implantation based on investigator's judgement;
7. A cooperative attitude to follow up the study procedures (Caregivers in case of minors).

Exclusion Criteria:

1. Known or suspected intolerances against anaesthesia;
2. Bad general condition (ECOG index >2);
3. Clinical and/or laboratory signs of acute systemic infections and/or severe inflammation at the time of screening. Patient can be re-screened after appropriate treatment;
4. Severe systemic disease (i.e. uncompensated diabetes);
5. Stenosis or retraction secondary to medical conditions other than hypospadias failure (i.e. radiotherapy, lichen sclerosis, etc…);
6. Allergy, sensitivity or intolerance to drugs or excipients (hypersensitivity to any of the excipients listed in Investigator's brochure or in this protocol):

   * Transport medium (Dulbecco's Modified Eagles Medium supplemented with L-glutamine)
   * Fibrin support;
7. Contraindications to the post- treatment local or systemic antibiotics and/or corticosteroids;
8. UTI or urine culture positive requiring a re-screening of patient;
9. Contraindications to undergo extensive surgical procedures;
10. Clinically significant or unstable concurrent disease or other clinical contraindications to stem cell implantation based on investigator's judegment or other concomitant medical conditions affecting grafting procedure;
11. Patients and parents/tutor unlikely to comply with the study protocol or unable to understand the nature and scope of the study or the possible benefits or unwanted effects of the study procedures and treatments;
12. Participation in another clinical trial where conventional investigational drug was received less than 1 months prior to screening visit;
13. Patients who received surgical procedure within 6 months prior to screening visit;
14. Anaesthesia or severe hypoesthesia of the area;
15. Diagnosis of local or systemic neoplastic disease.

Ages: 5 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients experiencing AESI | 3 months after treatment
  To demonstrate the safety of Holour in terms of AESI (persistent fever, infections)
Number and percentage of patients experiencing ADRs | 3 months after treatment
  To demonstrate the safety of Holour in terms of ADRs
Number and percentage of patients experiencing SAEs | 3 months after treatment
  To demonstrate the safety of Holour in terms of SAEs
Number and percentage of patients experiencing Serious ADRs | 3 months after treatment
  To demonstrate the safety of Holour in terms of Serious ADRs
Number and percentage of patients experiencing AESI | 12 months after treatment
  To demonstrate the safety of Holour in terms of AESI (persistent fever, infections)
Number and percentage of patients experiencing ADRs | 12 months after treatment
  To demonstrate the safety of Holour in terms of AESI ADRs
Number and percentage of patients experiencing SAEs | 12 months after treatment
  To demonstrate the safety of Holour in terms of SAEs
Number and percentage of patients experiencing Serious ADRs | 12 months after treatment
  To demonstrate the safety of Holour in terms of Serious ADRs
Number of patients with implantation success | 12 months after treatment
  Implantation success is defined on the basis of the degree of clinical (no lesions, no significant retractions) epithelial stability on the transplanted area. The degree of epithelial stability will be evaluated by visual inspection, cistouretrography, uretroscophy and checked for evaluating reepithelialization, erosions, infection, etc. and documented with photos with measures.
percentage of patients with implantation success | 12 months after treatment
  Implantation success is defined on the basis of the degree of clinical (no lesions, no significant retractions) epithelial stability on the transplanted area. The degree of epithelial stability will be evaluated by visual inspection, cistouretrography, uretroscophy and checked for evaluating reepithelialization, erosions, infection, etc. and documented with photos with measures.

SECONDARY OUTCOMES:
Number of patients with the treatment efficacy after Holour implantation and surgical reconstruction | up to 1 year after implantation
  Regeneration of a clinically normal appearing urethra epithelium with absence of detectable erosions/retractions and Clinical functionality (uroflowmetry) after the second step (urethral reconstruction) of transplant.
Evaluation of the percentage of re-epithelialization | up to 1 year after implantation
  Evaluation of the percentage of re-epithelialization
Evaluation of the clinical epithelial stability on the transplanted area by visual inspections | up to 1 year after implantation
  Evaluation of the regeneration of a clinically normal appearing epithelium with absence of detectable erosions/retractions
Evaluation of scar retraction presence | up to 1 year after implantation
  Evaluation of the penile retraction due to presence/absence of scars
Evaluation of uroflowmetry rate | From 3 to 12 months after the treatment
  Evaluation of the change of uroflowmetry compared to the baseline value with change of the curve shape and significant increase of the qmax flow rate;
Evaluation of the post-void residual volume through uroflowmetry | From 3 to 12 months after the treatment
  Evaluation of the change of the post-void residual compared to the baseline
Evaluation of the presence and severity of surgical complications | up to 1 year after implantation
  Presence and severity of surgical complications using the Clavien Dindo scale with the classification into 5 grades (I, II, III, IV and V from no need for clinical intervention to the death of the patient)
Evaluation of the adeverse events in terms of SAEs, AESI, ADR Serious ADRs, | up to 1 year after implantation
  Evaluation of the adeverse events in terms of SAEs, AESI, ADR Serious ADRs,

CONTACTS AND LOCATIONS:
Overall Officials: Graziella Pellegrini, Professor, Study Director — Holostem s.r.l.; Gianantonio Manzoni, MD, Principal Investigator — Fondazione IRCCS Cà Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Cà Granda, Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No